CLINICAL TRIAL: NCT02939105
Title: DualSculpting the Upper Arms Using Vacuum Applicators and a Customized Treatment Approach
Brief Title: CoolSculpting Treatment in the Upper Arms
Acronym: ARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA16-005
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CoolSculpting Treatment in the Upper Arm (Experimental): Subjects in the study were treated with the CoolSculpting System with one of two vacuum applicator types for bilateral fat reduction in the upper arms. Applicators were used concurrently, with an applicator on each arm. Each subject received 1 or 2 cooling cycles on each arm for 35 minutes at protocol-defined temperatures.
  The Investigator selected the applicator for each subject based on the intended fat volume of the treatment area.
  Interventions: Device: The ZELTIQ CoolSculpting System

INTERVENTIONS:
Device: The ZELTIQ CoolSculpting System — The CoolSculpting device will be used to perform treatments.

SUMMARY:
Evaluate the safety and efficacy of the ZELTIQ CoolSculpting System using specialized vacuum applicators for non-invasive subcutaneous fat reduction of the upper arms.

DETAILED DESCRIPTION:
Subcutaneous fat reduction of the upper arms using 2 vacuum applicator types will be done concurrently, such that a subject will have an applicator placed on each arm simultaneously.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 22 years of age and < 65 years of age.
* Subject has clearly visible fat sufficient for treatment on the upper arm, which in the investigator's opinion, may benefit from the treatment.
* No weight change exceeding 5% in the preceding month.
* Subject agrees to maintain his/her weight (i.e., within 5% of total body weight) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject has read and signed the study written informed consent form.

Exclusion Criteria

* History of a fat reduction procedure (e.g., liposuction, surgery, lipolytic agents, etc.), or implants in or adjacent to the area of intended treatment.
* History of prior surgery in the arms.
* Known history of cryoglobulinemia, cold urticaria, cold agglutinin disease, or paroxysmal cold hemoglobinuria.
* Known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* History of carpal tunnel syndrome, compartment syndrome or deep vein thrombosis in the upper extremities.
* Currently taking or has taken diet pills or weight control supplements within the past month.
* Any dermatological conditions, such as scars, infection, in the location of the treatment area that may interfere with the treatment or evaluation.
* Active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Pregnant or intending to become pregnant in the next 5 months.
* Lactating or has been lactating in the past 6 months.
* Unable or unwilling to comply with the study requirements.
* Currently enrolled in a clinical study of any other unapproved investigational drug or device. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rivers, MD, Principal Investigator — Pacific Dermaesthetics
Locations (1):
- Pacific Dermaesthetics, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rivers JK, Ulmer M, Vestvik B, Santos S. A customized approach for arm fat reduction using cryolipolysis. Lasers Surg Med. 2018 Mar 22. doi: 10.1002/lsm.22811. Online ahead of print. PMID 29566270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects seeking a reduction in upper arm fat were recruited from the general population.
Groups:
- CoolSculpting Intervention Group: The CoolSculpting System was used in the study. The study was designed to evaluate the safety and effectiveness of cryolypolysis for non-invasive reduction of upper arm fat.
Period: Overall Study
Arm/Group | CoolSculpting Intervention Group
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Fifteen subjects were enrolled and treated in the study.
Groups:
- CoolSculpting Intervention Group: Subjects treated with CoolSculpting System for Arm Fat
Arm/Group | CoolSculpting Intervention Group
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 51.1 [40 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 15
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 26.8 [22.4 to 33.7]
Fitzpatrick Skin Type [Number; unit: participants in skin type category] — The Fitzpatrick Skin Type scale is a numerical classification schema for human skin color, developed as a way to estimate the response of different skin types of skin to ultraviolet (UV) light. Fitzpatrick skin type characteristics are present at birth. The scales is composed of six skin type classifications for FST I to FST VI.
  There is no additional value in the skin type scale, e.g., a FST VI classification is no more or less valuable than a classification of FST I, FST II, FST III, FST IV or FST V.
  participants in skin type category
    FST I -always burns, never tans | 0
    FST II- burns easily, tans poorly | 9
    FST III- tans after initial burn | 4
    FST IV - burns minimally, tans easily | 0
    FST V- rarely burns, tans darkly easily | 2
    FST VI- never burns | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Correctly Identified Pre-treatment Photos
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images. Reviewers are practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images are presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. Criteria for evaluable photos for the purposes of the independent review: subject completed treatment regimen; subject has complete set of baseline photos; subject has a complete set of post-treatment photos; photos were taken using Zeltiq standard procedure. The expected success rate is 70% correct identification by 2 out of 3 reviewers.
Time Frame: 12 weeks post-final treatment
Population: The analysis population included subjects with baseline and post-treatment photos.
Measure: Count of Units; unit: photos
Units Other Than Participants: photos
Groups:
- CoolSculpting Intervention Group: Subjects treated with CoolSculpting for arm fat
Arm/Group | CoolSculpting Intervention Group
Number analyzed (Participants) | 15
Number analyzed (photos) | 30
photos | 26
Statistical Analysis 1: Comparison: CoolSculpting Intervention Group; Test type: Other; success proportion = 86.7, 95% CI 2-sided [69.3 to 96.2]

2. Primary Outcome: Number of Participants With Unanticipated Adverse Device Effects (UADE) Associated With the CoolSculpting System and Vacuum Applicators in the Upper Arms
Description: The primary safety endpoint of the study is the incidence of unanticipated adverse device effects (UADE) reported in the study period. Investigators assessed each adverse event to determine if there was relationship to the study device or procedure. Adverse event data are collected from the time of study enrollment through the final follow-up visit at 12 weeks post-treatment.
Time Frame: Enrollment through12 weeks post-final treatment
Population: Each adverse event occurring in the per-protocol population of 15 subjects was evaluated by investigators for any relationship to the study device or procedure.
Measure: Number; unit: number of participants with UADE
Arm/Group | CoolSculpting Intervention Group
Number analyzed (Participants) | 15
number of participants with UADE | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through the 12-week post-treatment follow-up visit.
Groups:
- CoolSculpting Intervention Group: CoolSculpting Treatment for Arm Fat
Arm/Group | CoolSculpting Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02939105/Prot_SAP_000.pdf